CLINICAL TRIAL: NCT04073290
Title: Prevention of Hepatic Encephalopathy by Administration of Rifaximin and Lactulose in Patients With Liver Cirrhosis Undergoing TIPS Placement: a Multi-centre Randomized, Double Blind, Placebo Controlled Trial.
Brief Title: Prevention of Post-TIPS Hepatic Encephalopathy by Administration of Rifaximin and Lactulose
Acronym: PEARL
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Erasmus Medical Center (Other); Leiden University Medical Center (Other); Maastricht University Medical Center (Other); Radboud University Medical Center (Other); University Medical Center Groningen (Other); Universitaire Ziekenhuizen KU Leuven (Other); Norgine (Industry)
Responsible Party: Principal Investigator, Dr. Bart Takkenberg, Study Chair, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PEARL trial; 2018-004323-37 (EudraCT Number); 848017009 (Other Grant/Funding Number: ZonMw)
Record Dates: First submitted 2019-08-27; First posted 2019-08-29 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Hepatic Encephalopathy; Cirrhosis, Liver; Portal Hypertension; Liver Diseases; Pathological Processes
Keywords: Rifaximin; Lactulose; post-TIPS HE; Prevention
MeSH Terms: conditions — Hepatic Encephalopathy; Liver Cirrhosis; Hypertension, Portal; Liver Diseases; Pathologic Processes | interventions — Rifaximin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rifaximin and lactulose (Active Comparator): Rifaximin 550 milligram b.i.d. combined with lactulose
  Interventions: Drug: Rifaximin 550 milligram Oral Tablet [XIFAXAN]; Drug: Lactulose 667 milligram/milliliter Oral Solution
- Placebo and lactulose (Placebo Comparator): Placebo b.i.d. combined with lactulose
  Interventions: Drug: Placebo oral tablet; Drug: Lactulose 667 milligram/milliliter Oral Solution

INTERVENTIONS:
Drug: Rifaximin 550 milligram Oral Tablet [XIFAXAN] — Rifaximin 550 milligram b.i.d. 72 hours before TIPS placement till 3 months post-TIPS
  Other Names: TARGAXAN
  Arms: Rifaximin and lactulose
Drug: Placebo oral tablet — Placebo b.i.d. 72 hours before TIPS placement till 3 months post-TIPS
  Other Names: Placebo
  Arms: Placebo and lactulose
Drug: Lactulose 667 milligram/milliliter Oral Solution — Lactulose based on soft stool frequency, 72 hours before TIPS placement till 3 months post-TIPS
  Other Names: Lactulose syrup

SUMMARY:
Rationale: Hepatic encephalopathy (HE) is a major and common complication in patients with liver cirrhosis. HE can be classified in the extensive range of neurocognitive deterioration as minimal HE (MHE), covert HE (grade I), or overt HE (OHE, grade II-IV). Liver cirrhosis is the most common cause of portal hypertension (PH). Patients who develop complications of PH, like variceal bleeding or refractory ascites, can benefit from a Transjugular Intrahepatic Portosystemic Shunt (TIPS) placement. Unfortunately, post-TIPS HE is a common and often severe complication. Incidence of new onset or worsening of HE after TIPS is approximately 20-45%. Currently there is no strategy to prevent post-TIPS HE.

DETAILED DESCRIPTION:
Objective: To assess the incidence of post-TIPS OHE within the first three months after prophylactic administration of lactulose and rifaximin versus placebo in patients who undergo Transjugular Intrahepatic Portosystemic Shunt (TIPS) placement.

Study design: A multicentre, randomized, placebo-controlled, double blind study.

Study population: Adult consecutive patients undergoing elective TIPS placement (for refractory ascites or secondary prophylaxis in variceal bleeding) in all Dutch academic centres where TIPS procedures are performed: Amsterdam UMC, location Academic Medical Centre (AMC), Erasmus MC, Leiden University Medical Centre (LUMC), Maastricht University Medical Centre+ (MUMC+), Radboud University Medical Centre (Radboudumc), University Medical Centre Groningen (UMCG), and University Hospitals Leuven (UZ Leuven) in Belgium.

Intervention: Rifaximin 550 milligram (mg) b.i.d. will be prescribed, in combination with a starting dose of 25 milliliter (mL) lactulose b.i.d. and further dependent on the amount of daily bowel movements, with the objective not to exceed more than two soft stools per day. Intervention will start 72 hours before TIPS placement, and will last till three months after TIPS placement. The control group will receive placebo in combination with lactulose (as described above).

Main study parameters/endpoints: Primary endpoint is the development of OHE within three months after TIPS placement determined by the West Haven criteria. Secondary endpoints are 90 day mortality; development of a second episode of OHE within the first three months; development of OHE in the period between three and twelve months after TIPS placement; development of MHE between TIPS placement and twelve months after placement; the increase of the psychometric hepatic encephalopathy score (PHES) and simplified one minute animal naming test (S-ANT1) compared to baseline. Differences in molecular composition of peripheral / portal blood samples at TIPS placement. Furthermore, quality of life will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Elective TIPS placement for refractory ascites or recurrent variceal bleeding:

   Recurrent tense ascites and one or more of the following criteria:

   i. Not responding to the maximal dose of diuretics (400 milligram spironolactone and 160 milligram furosemide).

   ii. Kidney insufficiency (Creatinine > 135 umol/L) induced by diuretics. iii. Electrolyte disturbances (Sodium < 125 mmol/L, Potassium > 5.5 mmol/L) induced by diuretics.

   iv. Not tolerating higher dose of diuretics (e.g. because of subjective side effects like muscle cramps).

   Recurrent variceal bleeding, not responsive to treatment with endoscopic band ligation and beta-blockers, with a high risk of failure of endoscopic treatment:

   i. Patients with a variceal bleeding and Child-Pugh C (10-13 points) cirrhosis or ii. Patients with a variceal bleeding, Child-Pugh B and an active bleeding during endoscopy
2. Age ≥18 years
3. Confirmed liver cirrhosis as documented by liver biopsy, elastography (e.g. Fibroscan) or combination of usual radiological and biochemical criteria.
4. Signed informed consent

Exclusion Criteria:

1. Any absolute contraindications for TIPS placement
2. Use of ciclosporin
3. Life-threatening variceal bleeding with emergency TIPS placement which can not be delayed 72 hours
4. Age > 80 years
5. Non-cirrhotic portal hypertension
6. Portal vein thrombosis (main trunk)
7. HIV
8. Current or recent (<3 months) use of rifaximin
9. Overt neurologic diseases such as Alzheimer's disease, Parkinson's disease
10. Pregnant or breastfeeding women
11. Patients refusing or unable to sign informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Estimated)
Dates: Start 2020-01-21 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
post-TIPS Hepatic Encephalopathy | First 3 months after TIPS placement
  post-TIPS Hepatic Encephalopathy

SECONDARY OUTCOMES:
Mortality | 90 days
  Mortality
Transplant free survival | One year
  Transplant free survival
time to development of post-TIPS HE episode(s) | One year
  time to development of post-TIPS HE episode(s)
development of a second episode of post-TIPS HE | 3 months
  development of a second episode of post-TIPS HE
development of post-TIPS HE between 3-12 months after TIPS placement | 3-12 months
  development of post-TIPS HE between 3-12 months after TIPS placement
change in Psychometric Hepatic Encephalopathy Score (PHES) compared to baseline | One year
  change in total PHES score compared to baseline (range -15 - +5) a lower score is a worse outcome
change in one-minute animal naming test compared to baseline | One year
  change in one-minute animal naming test compared to baseline
differences in molecular composition of peripheral / portal blood samples | One year
  differences in molecular composition of peripheral / portal blood samples at TIPS placement
differences in molecular composition of peripheral blood samples | One year
  differences in molecular composition of peripheral blood samples at baseline, compared to day 10 post-TIPS, week 4, week 12, and week 52;

OTHER OUTCOMES:
Health related Quality of life | One year
  Health related Quality of life, measured by EuroQol-5 Dimensions-5 Levels (EQ-5D-5L) questionnaire
Disease rrelated Quality of life | One year
  Health related Quality of life, Liver Disease Symptom Index (LDSI) 2.0 questionnaire.
Cost-effectiveness | One year
  Cost-effectiveness, measured by a combined questionnaire, based on institute for Medical Technology Assessment (iMTA) Productivity Cost Questionnaire (iPCQ)/Medical Consumption Questionnaire (iMCQ)

CONTACTS AND LOCATIONS:
Overall Officials: Bart Takkenberg, MD, PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (6):
- Universitaire Ziekenhuizen Leuven, Leuven, Belgium
- Netherlands (5):
  - Academic Medical Centre, Amsterdam
  - University Medical Center Groningen, Groningen
  - Leiden University Medical Center, Leiden
  - Radboud University, Nijmegen
  - Erasmus Medical Center, Rotterdam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zacharias HD, Kamel F, Tan J, Kimer N, Gluud LL, Morgan MY. Rifaximin for prevention and treatment of hepatic encephalopathy in people with cirrhosis. Cochrane Database Syst Rev. 2023 Jul 19;7(7):CD011585. doi: 10.1002/14651858.CD011585.pub2. PMID 37467180
- [Derived] de Wit K, Schaapman JJ, Nevens F, Verbeek J, Coenen S, Cuperus FJC, Kramer M, Tjwa ETTL, Mostafavi N, Dijkgraaf MGW, van Delden OM, Beuers UHW, Coenraad MJ, Takkenberg RB. Prevention of hepatic encephalopathy by administration of rifaximin and lactulose in patients with liver cirrhosis undergoing placement of a transjugular intrahepatic portosystemic shunt (TIPS): a multicentre randomised, double blind, placebo controlled trial (PEARL trial). BMJ Open Gastroenterol. 2020 Dec;7(1):e000531. doi: 10.1136/bmjgast-2020-000531. PMID 33372103